CLINICAL TRIAL: NCT03707275
Title: Personalized Voice Activated Wellness Assistants for Patients With Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medstar Health Research Institute (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Georgetown-Howard Universities Center for Clinical and Translational Science (Other); ObEN Artificial Intelligence (Unknown)
Responsible Party: Principal Investigator, Nawar Shara, Director, Department of Biostatistics and Biomedical Informatics, Medstar Health Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Alexa+ Study; UL1TR001409 (NIH)
Record Dates: First submitted 2018-10-02; First posted 2018-10-16 (Actual); Last update posted 2020-06-19 (Actual); Status verified 2020-06

CONDITIONS: Heart Failure; Congestive Heart Failure
Keywords: Clinical trial; Patient-centered outcomes; Treatment of heart failure; Technology in heart failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alexa+ Arm (Experimental)
  Interventions: Device: Alexa+
- Standard of Care Arm (Other)
  Interventions: Other: Standard of Care Arm

INTERVENTIONS:
Device: Alexa+ — Patients will receive the Amazon Echo Dot with Alexa voice technology (Alexa+) and will be asked to interact with the device for 3 months. Alexa+ will ask a series of questions. Based on the answers to these questions, it will either contact a study coordinator or will ask patients to take a specific action (such as weighing themselves). Data from this simple intervention will be merged with data extracted from the patient's health record and analyzed for clinical variables and demographics that are most predictive for success in use of these technologies.
  Arms: Alexa+ Arm
Other: Standard of Care Arm — This group will receive standard of care (SOC) HF management, which will entail regular follow up from the HF nurse and data from all hospital or clinic visits will be captured from the EHR.
  Arms: Standard of Care Arm

SUMMARY:
The Alexa+ Study will compare the use of the Amazon Echo Dot with Alexa voice technology in patients with chronic heart failure to those receiving standard of care heart failure management on changes in health and patient-centered outcomes.

DETAILED DESCRIPTION:
Integrating data from virtual voice activated assistants (Amazon Echo Dot with Alexa voice technology), with the rich medical history available in Electronic Health Records (EHR) will allow a truly customized, interactive, and automated personal healthcare assistant. This technology will be validated in patients who have chronic heart failure (HF). Half of the study patients will receive an Amazon Echo Dot (Alexa) enhanced with a HF Care custom Alexa Skill that is patient-specific, or Alexa+. Data on patient interactions with the device will be followed for three months. The control groups will receive standard of care (SOC) HF management. Both study and control groups will receive regular follow up from the HF nurse and data from all hospital or clinic visits will be captured from the EHR.

ELIGIBILITY:
Inclusion Criteria:

* Heart failure patients seen at the MedStar heart failure clinic and the MedStar Washington Hospital Center inpatient heart failure service
* At least 18 years of age
* Have access to in-home Wi-Fi

Exclusion Criteria:

* Participation in another interventional clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-12-10 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
Change in comfort level using Alexa+ technology as measured by the pre and post-test technology comfort survey | 3 months

SECONDARY OUTCOMES:
Change in number of hospitalizations as measured by hospitalization data extracted from the EHR | 3 months
Change in medication adherence as measured by number of prescriptions filled extracted from the EHR | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Nawar M Shara, M.S., PhD, Principal Investigator — Medstar Health Research Institute
Locations (1):
- MedStar Washington Hospital Center, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No
The findings from this study will be disseminated through formal presentations and informal frequent communications with participants in this study. Results will be presented at a national meeting and a report to document the results of the pre-and-post questionnaires as well as the data generated from Alexa will also be shared with researchers as appropriate.